CLINICAL TRIAL: NCT03743532
Title: A Needs Survey of Urban Day Shelter Users and Preliminary Evaluation of Alternative Approaches to Combustible Cigarette Cessation: The Exchange Project
Brief Title: E-Cigarettes and Financial Incentives to Promote Tobacco Harm Reduction Among Adults Accessing Shelter Services
Acronym: EXCHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10124
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cigarette Smoking
Keywords: Smoking cessation; Contingency management; Financial incentives; E-cigarettes; Homelessness
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation; Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- E-Cigarette Switching (EC) (Experimental): Participants were provided with an e-cigarette device and nicotine pods and advised to completely switch from combustible cigarettes to e-cigarettes. Although participants in the EC group did not earn incentives for combustible cigarette abstinence, they were yoked with a participant in the EC+FI group (described below), and they earned the same weekly incentive amount as their counterpart earned for combustible cigarette abstinence credited to a reloadable study credit card.
  Interventions: Behavioral: E-cigarette Switching
- E-Cigarette Switching + Financial Incentives (EC+FI) (Experimental): Participants assigned to the EC+FI group received ECs and pods and were instructed to switch from combustible cigarettes to e-cigarettes as described above for the EC group. Participants also earned escalating financial incentives for self-reported and carbon-monoxide-verified combustible cigarette abstinence via credits to a reloadable study credit card. Participants who reported combustible cigarette use and/or had a CO level >6 ppm did not earn incentives that week, but could earn incentives at the next visit with the incentive value reset to the starting value.
  Interventions: Behavioral: E-cigarette Switching; Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: E-cigarette Switching — Participants provided with e-cigarette device and nicotine pods and advised to switch from combustible cigarettes to e-cigarettes.
  Other Names: EC
Behavioral: Financial Incentives — Participants earned incentives for carbon monoxide-verified combustible cigarette abstinence.
  Other Names: FI
  Arms: E-Cigarette Switching + Financial Incentives (EC+FI)

SUMMARY:
This randomized controlled trial evaluated the feasibility and potential efficacy of 1) e-cigarette switching (EC) or 2) e-cigarette switching + financial incentives for combustible cigarette cessation (EC+FI)

DETAILED DESCRIPTION:
The current study examined the feasibility of e-cigarette switching and financial incentives contingent on combustible cigarette abstinence to promote combustible cigarette cessation among urban day shelter guests (N=60). A total of 60 adults who accessed the Homeless Alliance day shelter in Oklahoma City, OK were randomly assigned to 1 of 2 groups and followed weekly from 1 week prior to a scheduled EC switch date through 4 weeks post-switch date, with a final 8-week post-switch follow-up. The intervention groups were: 1) e-cigarette switching (EC) or 2) EC switching + small financial incentives for carbon monoxide (CO) verified combustible cigarette abstinence (FI + EC). The primary outcomes were self-reported combustible cigarette abstinence over the previous 7 days with carbon monoxide (CO)-verification at 4- and 8- weeks follow-up. Secondary outcomes included changes in CO from baseline, days of combustible cigarette smoking, and continued e-cigarette use. Other feasibility outcomes included study retention and perceptions of the intervention.

ELIGIBILITY:
1. ≥21 years of age
2. Expired CO level ≥8 ppm suggestive of current smoking
3. reported smoking ≥5 cigarettes per day
4. Willing and able to attend 8 study visits over a 10-week period
5. Interested in switching from CCs to ECs
6. Willing to abstain from smoking cannabis for the duration of the study
7. Able to speak and understand English
8. Demonstrated >6th grade English literacy by earning a score ≥4 on the Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF),
9. Able to read a 3-sentence selection from the consent form
10. Not pregnant, breastfeeding, or planning to become pregnant.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Homeless Alliance, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Boozary LK, Frank-Pearce SG, Alexander AC, Sifat MS, Kurien J, Waring JJC, Ehlke SJ, Businelle MS, Ahluwalia JS, Kendzor DE. Tobacco use characteristics, treatment preferences, and motivation to quit among adults accessing a day shelter in Oklahoma City. Drug Alcohol Depend Rep. 2022 Nov 5;5:100117. doi: 10.1016/j.dadr.2022.100117. eCollection 2022 Dec. PMID 36844157
- [Result] Sifat MS, Alexander AC, Businelle MS, Frank-Pearce SG, Boozary LK, Wagener TL, Ahluwalia JS, Kendzor DE. E-Cigarette switching and financial incentives to promote combustible cigarette cessation among adults accessing shelter services: A pilot study. Drug Alcohol Depend Rep. 2024 Nov 6;13:100295. doi: 10.1016/j.dadr.2024.100295. eCollection 2024 Dec. PMID 39764385

RESULTS

PARTICIPANT FLOW:
Groups:
- E-Cigarette Switching (EC): Participants will be asked to completely switch from cigarettes to e-cigarettes. They will receive an e-cigarette device and pods during the first 4 weeks following a scheduled switch date.
  E-cigarette: Participants will receive an e-cigarette device and pods. Each participant in this group will be yoked to a participant in the financial incentives group, thus receiving equal payments. Yoking will reduce or eliminate differential attendance rates between groups because participants have the opportunity to earn the same amount of money regardless of group assignment. Participants will be followed for the first 4 weeks following a scheduled quit attempt.
- Financial Incentives + E-cigarette Switching: Participants will be asked to completely switch from cigarettes to e-cigarettes, and they will receive an e-cigarette device and pods during the first 4 weeks following a scheduled switch date. Participants will also receive weekly financial incentives for biochemically-verified cigarette abstinence during the first 4 weeks following the switch date.
  Financial incentives + E-cigarette: Participants will receive an e-cigarette device and pods and the opportunity to earn financial incentives for biochemically-verified cigarette smoking abstinence, credited to a gift card with biochemical evidence of smoking abstinence during the first 4 weeks following a scheduled quit attempt.
Period: Overall Study
Arm/Group | E-Cigarette Switching (EC) | Financial Incentives + E-cigarette Switching
Started | 30 | 30
Completed | 14 | 13
Not Completed | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- E-cigarette Switching + Financial Incentives (EC+FI): Participants will be asked to completely switch from cigarettes to e-cigarettes, and they will receive an e-cigarette device and pods during the first 4 weeks following a scheduled switch date. Participants will also receive weekly financial incentives for biochemically-verified cigarette abstinence during the first 4 weeks following the switch date.
  Financial incentives + E-cigarette: Participants will receive an e-cigarette device and pods and the opportunity to earn financial incentives for biochemically-verified cigarette smoking abstinence, credited to a gift card with biochemical evidence of smoking abstinence during the first 4 weeks following a scheduled quit attempt.
- Total: Total of all reporting groups
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching + Financial Incentives (EC+FI) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.30 (10.98) | 47.23 (10.94) | 48.77 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 30 | 26 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 13 | 20
  White | 19 | 13 | 32
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Currently Experiencing Homelessness [Count of Participants; unit: Participants] | 24 | 22 | 46
Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: Number of cigarettes smoked per day] — Population: 1 participant excluded from analyses because of out of range value (i.e., 2400 cigarettes per day).
  Number of cigarettes smoked per day
    number analyzed (Participants) | 30 | 29 | 59
    (all) | 15.73 (12.13) | 16.28 (11.08) | 16.00 (11.53)

OUTCOME MEASURES:

1. Primary Outcome: Combustible Cigarette Cessation
Description: Self-reported and Carbon monoxide-verified (<=6 ppm) combustible cigarette smoking abstinence during the previous 7 days (missing = smoking)
Time Frame: 4 weeks post-switch date
Population: Participants with missing cigarette smoking status were considered smoking.
Measure: Count of Participants; unit: Participants
Groups:
- E-cigarette Switching (EC) + Financial Incentives: Participants will be asked to completely switch from cigarettes to e-cigarettes, and they will receive an e-cigarette device and pods during the first 4 weeks following a scheduled switch date. Participants will also receive weekly financial incentives for biochemically-verified cigarette abstinence during the first 4 weeks following the switch date.
  Financial incentives + E-cigarette: Participants will receive an e-cigarette device and pods and the opportunity to earn financial incentives for biochemically-verified cigarette smoking abstinence, credited to a gift card with biochemical evidence of smoking abstinence during the first 4 weeks following a scheduled quit attempt.
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 30 | 30
Participants | 1 | 4

2. Primary Outcome: Combustible Cigarette Cessation
Description: as for outcome 1
Time Frame: 8 weeks post-quit/switch date
Population: Participants with missing cigarette smoking status were considered smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching + Financial Incentives (EC+FI)
Number analyzed (Participants) | 30 | 30
Participants | 3 | 4

3. Secondary Outcome: Combustible Cigarette Cessation (Complete Case Analysis)
Description: Self-reported and Carbon monoxide-verified (<=6 ppm) combustible cigarette smoking abstinence during the previous 7 days (missing excluded)
Time Frame: 4 weeks post-switch
Population: Participants with missing smoking status were excluded from the analyses (i.e., complete case analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 16 | 15
Participants | 1 | 4

4. Secondary Outcome: Combustible Cigarette Cessation (Complete Case Analysis)
Description: as for outcome 3
Time Frame: 8 weeks post-switch
Population: Participants with missing smoking status data were excluded from the analyses (i.e., complete case analysis).
Measure: Count of Participants; unit: Participants
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 14 | 13
Participants | 3 | 4

5. Secondary Outcome: Expired Carbon Monoxide (CO), Parts Per Million (Ppm), Change From Baseline
Description: Change in expired CO (ppm) from baseline to 4 weeks post-switch-date.
Time Frame: 4 weeks post-switch
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 16 | 15
ppm | 0.31 (12.10) | -8.73 (7.77)

6. Secondary Outcome: Expired Carbon Monoxide (CO), Parts Per Million (Ppm), Change From Baseline
Description: Change in expired CO (ppm) from baseline to 8 weeks post-switch-date
Time Frame: 8 week post-switch
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 14 | 13
ppm | -4.57 (8.91) | -7.23 (9.35)

7. Secondary Outcome: Days of Combustible Cigarette Smoking, Past 7 Days
Description: The total number of days of combustible cigarette smoking during the past week
Time Frame: 4 weeks post-switch
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 16 | 15
Days | 4.25 (2.77) | 2.20 (2.60)

8. Secondary Outcome: Days of Combustible Cigarette Smoking, Past 7 Days
Description: The total number of days of combustible cigarette smoking during the past 7 days
Time Frame: 8 weeks post-switch
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 14 | 11
Days | 2.79 (2.33) | 3.73 (3.32)

9. Secondary Outcome: Days of E-cigarette Use, Past 7 Days
Description: The total number of days where e-cigarettes were used during the past 7 days
Time Frame: 4 weeks post-switch
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 14 | 14
Days | 3.64 (2.84) | 5.07 (2.84)

10. Secondary Outcome: Days of E-cigarette Use, Past 7 Days
Description: The total number of days on which E-cigarettes were used during the past 7 days
Time Frame: 8 weeks post-switch
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
Number analyzed (Participants) | 13 | 11
Days | 4.15 (3.11) | 4.18 (3.25)

11. Secondary Outcome: Follow-Up Completion
Description: The number of participants who completed the smoking status follow-up assessment.
Time Frame: 4 weeks post-switch
Measure: Count of Participants; unit: Participants
Arm/Group | E-Cigarette Switching (EC) | E-Cigarette Switching + Financial Incentives (EC+FI)
Number analyzed (Participants) | 30 | 30
Participants | 16 | 15

12. Secondary Outcome: Follow-Up Completion
Description: The number of participants who completed the smoking status follow-up assessment
Time Frame: 8 weeks post-switch
Measure: Count of Participants; unit: Participants
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching + Financial Incentives (EC+FI)
Number analyzed (Participants) | 30 | 30
Participants | 14 | 13

ADVERSE EVENTS:
Time Frame: Approximately 10 weeks
Arm/Group | E-Cigarette Switching (EC) | E-cigarette Switching (EC) + Financial Incentives
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03743532/Prot_SAP_000.pdf